CLINICAL TRIAL: NCT03435237
Title: Phenotyping Asthma for Bronchial Thermoplasty: Airway Smooth Muscle Structure and Function
Brief Title: Phenotyping Asthma for Bronchial Thermoplasty
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melissa J. Suter, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2017P000962; 1R01HL133664-01A1 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2018-02-15 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Severe Asthma
Keywords: Optical Coherence Tomography; Bronchial Thermoplasty
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage samples will be taken before and after the completion of the bronchial thermoplasty procedure to determine inflammation level of the lung.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate a new imaging technology, called optical coherence tomography (OCT) to examine the asthmatic airways before and after bronchial thermoplasty, which is a new treatment option for severe asthmatic patients. The aim of this study is to learn more about how airways respond to this new treatment. In the future the investigators hope OCT will aid clinicians in the initial assessment, management and long-term follow up of patients receiving bronchial thermoplasty.

DETAILED DESCRIPTION:
Asthma currently affects over 300 million individuals worldwide and the number of the affected patient is continuously increasing. Approximately 10% of asthmatics have poorly controlled, severe symptoms.

The exact mechanisms behind the development of asthma are unknown. However, the excessive contraction of airway smooth muscle leading to airway constriction is thought to be responsible for the majority of the symptoms of asthma. A new treatment option, termed bronchial thermoplasty, can offer relief for individuals with severe asthma. Bronchial thermoplasty works by reducing smooth muscle with thermal energy.

This new imaging technology, called optical coherence tomography (OCT) is the first imaging modality that is capable to visualize airway smooth muscle in humans. In this study the investigators will examine the asthmatic airways before and after bronchial thermoplasty to learn about how airways respond to this treatment. The long term goal of this study is to use OCT to look at the airways with the hope of helping clinicians monitor and predict the response to bronchial thermoplasty.

During the scheduled bronchial thermoplasty procedure, OCT imaging will be performed. The study imaging will add less than 10 minutes to the time required for the standard procedure.Twelve months following the completion of bronchial thermoplasty, the investigators will ask the participants to return to the hospital to undergo follow-up tests including a CT scan and a bronchoscopy procedure with repeat OCT imaging. The investigators expect these test to be accomplished in 2 additional visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing elective bronchial thermoplasty
2. Patient is between the ages of 18 and 60
3. Patient is able to give informed consent
4. Negative pregnancy test for all female of childbearing potential who are sexually active and not using contraception, are seeking to become pregnant, or who are nursing.
5. Nonsmoking (<5 pack year tobacco exposure)
6. No history of co-existing lung disease
7. Meet American Thoracic Society criteria for diagnosis of asthma with either/or

   1. Bronchodilator response to albuterol (≥12% change in FEV1)
   2. Positive methacholine bronchoprovocation (PC20 < 25 mg/ml)

Exclusion Criteria:

1. Patients who are pregnant.
2. Patient does not meet the requirements to undergo clinical bronchial thermoplasty, as determined by the treating physician

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients referred to the Division of Pulmonary and Critical Care Medicine at Massachusetts General Hospital or Beth Israel Deaconess Medical Center for bronchial thermoplasty for the treatment of uncontrolled asthma will be eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate OCT for assessing bronchial thermoplasty | 1 year
  Does OCT imaging detect biomarkers that may predict patient's clinical response to bronchial thermoplasty as assessed by the Asthma Quality of Life Questionnaire.
Evaluate OCT for assessing bronchial thermoplasty | 1 year
  Does OCT imaging detect biomarkers that may predict patient's clinical response to bronchial thermoplasty as assessed by the pulmonary function tests.
Evaluate OCT for assessing bronchial thermoplasty | 1 year
  Does OCT imaging detect biomarkers that may predict patient's clinical response to bronchial thermoplasty as assessed by airway inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Suter, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No